CLINICAL TRIAL: NCT05571709
Title: Does an Acute Exercise Bout Increases Soluble and Muscle Myokine Concentration in Healthy, Older Persons
Brief Title: The Effect of Exercise on Myokine Production in Aging Persons
Acronym: EXI-AGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Niels Hellings, Professor Doctor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: B1152022000006
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Aging; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Aged individuals who perform exercise training are compared to aged individuals who remain sedentary.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aged individuals who perform exercise training (Active Comparator): Aged individuals will perform an acute bout of resistance trainig (30 minutes). This training is focused on the lower limbs.
  Interventions: Other: Exercise training; Behavioral: Questionnaire; Procedure: Percutaneous muscle biopsy; Procedure: Blood sample
- Aged individuals who stay sedentary (Sham Comparator): Aged individuals will remain seated for 30 minutes.
  Interventions: Behavioral: Questionnaire; Procedure: Percutaneous muscle biopsy; Procedure: Blood sample

INTERVENTIONS:
Other: Exercise training — Resistance training of the lower limbs
  Arms: Aged individuals who perform exercise training
Behavioral: Questionnaire — Physical activity questionnaire
Procedure: Percutaneous muscle biopsy — Muscle biopsy of the vastus lateralis (m. quadriceps)
Procedure: Blood sample — Venous blood sample

SUMMARY:
The incidence of age-related diseases, such as cancer and cardiovascular diseases, rapidly rises. These days, age-related diseases cause the majority of all healthcare expenses. During ageing senescent cells secrete a range of harmful inflammatory signals, which leads to chronic inflammation (inflamm-aging) and accelerates aging throughout the rest of the body. Interestingly, people who regularly exercise show less signs of inflamm-aging compared to people with a sedentary lifestyle. Molecules secreted by skeletal muscles, called myokines, may play an important role. However, the underlying molecular mechanisms remain unknown. This pilot study aims to investigate if an acute bout of resistance training is an appropriate tool to induce an increase in the release of muscle derived myokines in aged persons.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons

Exclusion Criteria:

* Smoking
* Infection < 2 weeks ago
* Received a vaccine < 2 weeks ago
* Allergy to Lidocain
* Immune deficiency
* Presence of a tumour or in treatment
* Usage of anti-coagulant medication
* Presence of following conditions:

  * Haemophilia
  * Auto-immune disease
  * Cardiovascular disease
  * Musculoskeletal diseases which refrains the patient from exercising

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cytokine concentration | Day 2
  Measurement of multiple cytokines in blood (for example: IL-6, IL-15, IL-4, irisin...) with ELISA's or multiplex assays
Myokine production | Day 2
  Immunohistochemistry staining (fluorescent) of multiple myokines (for example: IL-6, IL-15, IL-4, irisin..) and aging markers (p16,p21...) on muscle tissue
Immune parameters | Day 2
  Flow cytometry panels of immune parameters in muscle tissue
Myokine protein levels | Day 2
  Western blotting of multiple myokines in muscle tissue
Myokine gene expression | Day 2
  Quantitative PCR (polymerase chain reaction) of markers in muscle tissue

SECONDARY OUTCOMES:
Blood pressure | Day 1
  The force of circulating blood on the walls of the arteries. Measured using an electronic sphygmomanometer
Resting Heart Rate | Day 1
  Measured using an electronic sphygmomanometer
International Physical Activity Questionnaire (Short form) | Day 1
  Measures the subjective level of activity of the last seven days. 7 questions regarding amount of time spent on certain activities.

CONTACTS AND LOCATIONS:
Overall Officials: Chiel Hex, MD., Principal Investigator — University of Hasselt
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No